CLINICAL TRIAL: NCT04640844
Title: Contribution of the Pharmacological Profile of the A2A Receptor to Adenosine in the Diagnosis of Myocardial Ischemia
Acronym: RIMACI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-13; 2020-A00686-33 (Other: idrcb)
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Chronic Coronary Artery Disease
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients hospitalized (Experimental): for surgery of the aorta and / or arteries of the lower limbs.
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — measuring the expression and function of lymphocyte A2A receptors.

SUMMARY:
The chronic coronary artery disease could be detected by a drop in the expression of A2A receptors to adenosine, while high values of the KD / EC50 ratio are a sign of coronary ischemia. Knowing the number of A2A receptors in circulating lymphocytes could allow detection of coronary artery disease and evaluating the functionality of A2A receptors in circulating lymphocytes could allow quantification of myocardial ischemia.

Thus, a simple and unique blood sample would quickly detect patients with life-threatening coronary ischemia. This would avoid prolonged hospitalizations and costly non-invasive tests (stress echocardiography, myocardial scintigraphy) in patients without coronary artery disease.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the discriminating capacities of A2A adenosine receptors expression on the surface of circulating lymphocytes for the detection of coronary artery disease in patients hospitalized for surgery of the aorta and / or arteries of the lower limbs.

The secondary objectives are:

Assessment of the discriminating capacities of the functionality (KD / EC50) of A2A adenosine receptors on the surface of circulating lymphocytes, for the diagnosis of myocardial ischemia in patients hospitalized for surgery of the aorta and / or arteries of legs.

Determinate the best threshold for discriminating patients with coronary artery disease and estimate the discriminating performance associated with this threshold.

Determinate the best threshold for discriminating patients with myocardial ischemia and estimate the discriminating performance associated with this threshold.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for preoperative assessment of vascular surgery of the aorta and / or arteries of the lower limbs.
* Adult person (age> 18).
* Affiliated with a social security scheme.
* Signature of informed consent.

Exclusion Criteria:

* Patients with a history of coronary artery disease awaiting revascularization.
* Hyperthyroidism, anemia (Hb <13 g / dL).
* Contraindication to the practice of coronary angiography, stress echocardiography or myocardial scintigraphy.
* Unstable hemodynamic state or cardiogenic shock.
* Adults protected under guardianship, curatorship or legal protection.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dosage of adenosine | 24 MONTHS
  measuring the expression and function of lymphocyte A2A receptors.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO PRADALIE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France